CLINICAL TRIAL: NCT04308785
Title: A Multicenter, Double-Blind, Placebo-Controlled, Randomized, Phase 2 Study to Investigate the Efficacy and Safety of Atezolizumab With or Without Tiragolumab as Consolidation Therapy in Patients With Limited Stage Small Cell Lung Cancer Who Have Not Progressed After Chemoradiotherapy
Brief Title: A Study of Atezolizumab With or Without Tiragolumab Consolidation in Limited Stage Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The sponsor's decision was based on the negative results of SKYSCRAPER-02.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ML41257
Record Dates: First submitted 2020-03-12; First posted 2020-03-16 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Carcinoma, Small Cell Lung
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — atezolizumab; Tiragolumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Atezolizumab + Tiragolumab (Experimental): Participants will receive atezolizumab + tiragolumab intravenously on the first day of each cycle. One cycle of therapy will be defined as 21 days. Atezolizumab and tiragolumab treatment will continue up to 17 doses unless investigator-assessed loss of clinical benefit, unacceptable toxicity, investigator or patient decision to withdraw from therapy, or death (whichever occurs first).
  Interventions: Drug: Atezolizumab; Drug: Tiragolumab
- Arm B: Atezolizumab + Placebo (Experimental): Participants will receive atezolizumab + placebo on the first day of each cycle. One cycle of therapy will be defined as 21 days. Atezolizumab and placebo treatment will continue up to 17 doses unless investigator-assessed loss of clinical benefit, unacceptable toxicity, investigator or patient decision to withdraw from therapy, or death (whichever occurs first).
  Interventions: Drug: Atezolizumab; Other: Placebo

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered at a dose of 1200 mg intravenously on the first day of each 21-day cycle.
  Other Names: Tecentriq
Drug: Tiragolumab — Tiragolumab will be administered at a dose of 600 mg intravenously on the first day of each 21-day cycle.
  Arms: Arm A: Atezolizumab + Tiragolumab
Other: Placebo — Placebo matching to tiragolumab will be administered at a dose of 600 mg intravenously on the first day of each cycle.
  Arms: Arm B: Atezolizumab + Placebo

SUMMARY:
This is a multicenter, double-blind, placebo-controlled, randomized, phase II study to investigate the efficacy and safety of Atezolizumab with or without Tiragolumab as consolidation therapy in participants with limited stage small cell lung cancer who have not progressed during/after chemoradiotherapy.

DETAILED DESCRIPTION:
Participants can receive concurrent or sequential chemoradiotherapy (CRT) as per local standard of care, but they must be randomized within 6 weeks from completion of chemoradiotherapy. Participants should receive 4 cycles of chemotherapy and radiotherapy dose of 56-64 Gy (once daily) before randomization, and those participants who have not progressed during/after CRT will be stratified by response to CRT, radiotherapy timing, and be randomized in a 1:1 ratio to Atezolizumab+Tiragolumab arm or Atezolizumab+placebo arm.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* ECOG performance status of 0 or 1
* Histologically confirmed limited-stage SCLC.
* Patients who have not progressed during/after chemoradiotherapy.
* Concurrent or sequential chemoradiotherapy per local clinical practice must have been completed within 6 weeks prior to the first study treatment. If concurrent CRT is used, at least two cycles of chemotherapy should have been conducted during radiotherapy. If sequential radiotherapy is used, induction chemotherapy should be given 2 cycles of chemotherapy before thoracic radiotherapy.
* Adequate hematologic and end organ function.
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 5 months after the final dose of atezolizumab or placebo, and 90 days after the final dose of tiragolumab or placebo, and 6 months for chemotherapy after the last dose of chemotherapy treatment, whichever is later.
* For men: agreement to remain abstinent or use contraceptive measures and agreement to refrain from donating sperm.
* Patients must have recovered from all acute toxicities from previous therapy, excluding alopecia and toxicities related to prior therapy.
* Patients must submit a pre-treatment tumor tissue sample.

Exclusion Criteria:

* Histology mixtured or Extensive-stage SCLC (per the Veterans Administration Lung Study Group (VALG) staging system).
* Uncontrolled pleural effusion or pericardial effusion requiring recurrent drainage procedures
* Evidence of significant uncontrolled concomitant disease that could affect compliance with the protocol, including significant liver disease
* Malignancies other than SCLC within 5 years prior to study treatment initiation, with the exception of those with a negligible risk of metastasis or death treated with expected curative outcome
* Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or within 5 months after the final dose of atezolizumab and 90 days after the final dose of tiragolumab, and 6 months for chemotherapy after the final dose of the chemotherapy treatment.
* Active or history of autoimmune disease or immune deficiency
* Uncontrolled or symptomatic hypercalcemia
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.
* Positive test result for HIV
* Patients with active hepatitis B or hepatitis C virus
* Active tuberculosis
* Severe infections within 4 weeks prior to study treatment initiation, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
* Significant cardiovascular disease
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, anti-CTLA4, anti-tigit, anti-PD-1, and anti-PD-L1 therapeutic antibodies
* Unresolved toxic effects of grade 2 or higher (CTCAE 5.0), including grade ≥ 2 pneumonitis from previous therapy
* Active EBV infection or known or suspected chronic active EBV infection at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Investigator Assessed Progression-Free Survival (PFS) in the Intent-To-Treat (ITT) Population | Randomization up to approximately 48 months
  PFS is defined as the time from randomization to the first occurrence of disease progression or death from any cause, whichever occurs first. PFS will be calculated based on disease status evaluated by the investigator according to RECIST v1.1.

SECONDARY OUTCOMES:
Overall Survival (OS) in the ITT Population | Randomization up to approximately 48 months
  OS is defined as the time from randomization to death from any cause or last follow-up.
PFS Rate at 1 Year and 2 Years in the ITT Ppulation | Baseline to 1 Year and 2 Years
  PFS rate at 1 year and 2 years, defined as the proportion of patients remaining stable disease or ongoing response per RECIST v1.1 at 1 year and 2 years from the time of randomization.
OS Rate at 1 Year, 2 Years and 3 Years in the ITT Population | Baseline to 1 Year, 2 Years and 3 Years
  OS rate at 1 year, 2 years and 3 years is defined as the proportion of patients remaining alive 1 year, 2 years and 3 years from the time of randomization.
Objective Response Rate (ORR) in the ITT Population | Randomization up to approximately 48 months
  ORR is defined as the percentage of patients who attain complete response (CR) or partial response (PR) according to RECIST v1.1 in patients who have measurable disease at baseline.
Duration of Response (DOR) in the ITT Population | Time from first documentation of complete response (CR) or partial response (PR) up to approximately 48 months
  DOR is defined as the time interval from first occurrence of a documented objective response to the time of disease progression as determined by the investigator according to the RECIST v1.1 or death from any cause, whichever occurs first, in the patients who have experienced a CR or PR (unconfirmed) during the study.
Investigator Accessed Progression-Free Survival (PFS) in the Intent-To-Treat (ITT) Population by Response to Chemoradiotherapy (CRT) [Stable Disease (SD) vs. Complete Response (CR)/Partial Response (PR)] | Randomization up to approximately 33 months
  PFS is defined as the time from randomization to the first occurrence of disease progression or death from any cause, whichever occurs first. PFS will be calculated based on disease status evaluated by the investigator according to RECIST v1.1.
Overall Survival (OS) in the ITT Population by Response to CRT (SD vs. CR/PR) | Randomization up to approximately 48 months
  OS is defined as the time from randomization to death from any cause or last follow-up.
Objective Response Rate (ORR) in the ITT Population by Response to CRT (SD vs. CR/PR) | Randomization up to approximately 48 months
  ORR is defined as the percentage of patients who attain complete response (CR) or partial response (PR) according to RECIST v1.1.
Investigator Accessed Progression-Free Survival (PFS) in the Intent-To-Treat (ITT) Population by Radiotherapy Timing (Concurrent vs. Sequential) | Randomization up to approximately 48 months
  PFS is defined as the time from randomization to the first occurrence of disease progression or death from any cause, whichever occurs first. PFS will be calculated based on disease status evaluated by the investigator according to RECIST v1.1.
Overall Survival (OS) in the ITT Population by Radiotherapy Timing (Concurrent vs. Sequential) | Randomization up to approximately 48 months
  OS is defined as the time from randomization to death from any cause or last follow-up.
Objective Response Rate (ORR) in the ITT Population by Radiotherapy Timing (Concurrent vs. Sequential) | Randomization up to approximately 48 months
  ORR is defined as the percentage of patients who attain complete response (CR) or partial response (PR) according to RECIST v1.1.
Percentage of Participants With All Adverse Events Related to Atezolizumab and Atezolizumab + Tiragolumab Treatment in the ITT Population | Baseline up to approximately 48 months
Percentage of Participants With Serious and Non-Serious Immune Mediated Adverse Events Related to Atezolizumab and Atezolizumab + Tiragolumab Treatment in the ITT Population | Baseline up to approximately 48 months
Percentage of Participants With All Adverse Events Related to Treatment in the ITT Population | Baseline up to approximately 48 months
Time to Deterioration (TTD) in Patient-Rported Lung Cancer Symptoms | Randomization up to approximately 48 months
  TTD is defined as the time from randomization to a patient's first ≥10-point score change from baseline in a scale maintained for at least two consecutive PRO assessments, or followed by death within 3 weeks of the first ≥10-point score change.
EORTC QLQ-C30 Score | Day 1 of first 3 cycles (each cycle is 21 days) then with tumor assessments & 3 months after radiographic disease progression or for patients who continue atezolizumab after radiographic disease progression loss of clinical benefit up to approx 48 months
  EORTC QLQ-C30, European Organisation for Research and Treatment of Cancer Quality-of-Life Questionnaire-Core 30 Questionnaire, is a validated, reliable self-report measure. It consists of 30 questions that assess five aspects of patient functioning (physical, emotional, role, cognitive, and social), three symptom scales (fatigue, nausea and vomiting, pain), global health/quality of life, and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties) with a recall period of the previous week. Scale scores can be obtained for the multi-item scales.
EORTC QLQ-LC13 Score | Day 1 of first 3 cycles (cycle length=21 days), then with tumor assessments & 3 months after radiographic disease progression or for patients who continue atezolizumab after radiographic disease progression loss of clinical benefit up to approx 48 months
  The EORTC, European Organisation for Research and Treatment of Cancer Quality-of-Life Questionnaire, QLQ-LC13 is a modular supplement to the EORTC quality-of-life questionnaire for use in lung cancer. This module incorporates one multiple-item scale to assess dyspnea and a series of single items assessing pain, coughing, sore mouth, dysphagia, peripheral neuropathy, alopecia, and hemoptysis.
EuroQol 5-Dimension 5-Level (EQ-5D-5L) Index Based and Visual Analogue Scale (VAS) Scores | Day 1 of first 3 cycles (each cycle is 21 days) then with tumor assessments & 3 months after radiographic disease progression or for patients who continue atezolizumab after radiographic disease progression loss of clinical benefit up to approx 48 months
  The EuroQol 5-Dimension Questionnaire, 5-level version (EQ-5D-5L), is a validated self-report health status questionnaire that is used to calculate a health status utility score for use in health economic analyses. There are two components to the EQ-5D-5L: a five-item health state profile that assesses mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, as well as a visual analogue scale (VAS) that measures health state. Published weighting systems allow for creation of a single composite score of the patient's health status.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (17):
- China (17):
  - Beijing Cancer Hospital, Beijing
  - Jilin Cancer Hospital, Changchun
  - Hu Nan Provincial Cancer Hospital, Changsha
  - Sichuan Cancer Hospital, Chengdu
  - Southwest Hospital , Third Military Medical University, Chongqing
  - Fujian Cancer Hospital, Fuzhou
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Sun Yet-sen University Cancer Center, Guangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Anhui Province Cancer Hospital, Hefei
  - Shandong Cancer Hospital, Jinan
  - Guangxi Cancer Hospital of Guangxi Medical University, Nanning
  - Fudan University Shanghai Cancer Center; Medical Oncology, Shanghai
  - Tianjin Cancer Hospital, Tianjin
  - Tumor Center,Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - First Affiliated Hospital of Medical College of Xi'an Jiaotong University, Xi'an
  - Henan Cancer Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.clinicalstudydatarequest.com). Further details on Roche's criteria for eligible studies are available here (https://clinicalstudydatarequest.com/Study-Sponsors/Study-Sponsors-Roche.aspx). For further details on Roche's Global Policy on Sharing of Clinical Study Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).